CLINICAL TRIAL: NCT05147571
Title: RNS® System Responsive Thalamic Stimulation for Primary Generalized Seizures (NAUTILUS) Study
Brief Title: RNS System NAUTILUS Study
Acronym: NAUTILUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP10016
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy; Idiopathic Generalized Epilepsy; Generalized Tonic Clonic Seizure
Keywords: Medically refractory; Responsive neurostimulation; RNS System; Thalamic stimulation
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized; Epilepsy, Tonic-Clonic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Group (responsive stimulation ON) (Active Comparator): Participants are implanted with the RNS System and are receiving treatment with responsive stimulation.
  Interventions: Device: Responsive stimulation
- Sham Group (responsive stimulation OFF) (Sham Comparator): Participants are implanted with the RNS System and are not receiving treatment with responsive stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Responsive stimulation — The RNS System provides closed loop responsive brain stimulation. The Neurostimulator monitors the electrical activity of the brain to detect abnormal activity that could lead to a seizure. If abnormal activity is detected, the neurostimulator delivers electrical stimulation to the brain through the leads to help prevent the seizure before it occurs.
  Arms: Active Group (responsive stimulation ON)
Device: Sham stimulation — For those in the Sham Stimulation group, the RNS System will be set to detect abnormal activity but will not have responsive stimulation enabled. Both Sham and Active groups will undergo therapy testing at each appointment in order to maintain the blind.
  Arms: Sham Group (responsive stimulation OFF)

SUMMARY:
To demonstrate that the RNS System for thalamic stimulation is safe and effective as an adjunctive therapy for the reduction of primary generalized seizures in individuals 12 years of age or older who have drug-resistant idiopathic generalized epilepsy.

DETAILED DESCRIPTION:
NeuroPace is sponsoring the NAUTILUS Study with the RNS System for thalamic stimulation as an adjunctive therapy for the treatment of generalized seizures in individuals 12 years of age or older who have drug-resistant idiopathic generalized epilepsy. The RNS System is currently approved by the FDA for use in patients 18 years and older with hard-to-treat partial-onset seizures. The same device will be used in the NAUTILUS Study.

The study is a prospective, multicenter, single-blind, randomized, sham stimulation controlled pivotal study and participants will be followed for two years after placement of the RNS System. The study will enroll a maximum of 100 participants within the United States to ensure that at least 80 participants are implanted with the RNS System.

The study design includes a two-month retrospective and one-month prospective baseline. All participants will have detection enabled at the time of implant. At one month post-implant, participants will be randomized 1:1 to Active or Sham stimulation. For those randomized to the Active group, stimulation will be enabled. Participants will be blinded to their own randomization status until the 2nd GTC occurs for that individual, they completed the 9-month Effectiveness Evaluation Period (12-months post-implant), or the 60th GTC-event occurs in the group, whichever occurs first. After that, patients will be unblinded and patients in the Sham group (responsive stimulation OFF) will have responsive stimulation enabled (responsive stimulation ON).

ELIGIBILITY:
Inclusion Criteria:

* Participant is age 12 and older.
* Participant is male or is a female of childbearing potential who is surgically sterile, 2 years postmenopausal, or practices a reliable method of contraception (hormonal, barrier method or abstention).
* Participant failed treatment with a minimum of two antiseizure medications (used in appropriate doses) with adequate monitoring of compliance and the effects of treatment, as determined by the investigator.
* Participant is able to maintain an electronic diary alone or with the assistance of a competent individual.
* Participant is able to attend clinic appointments in accordance with the study schedule.
* Participant or parent(s) or legal representative have signed an IRB approved written informed consent/assent. The informed consent form or specific assent form, where required, will be signed and dated by minors.
* Participant is not currently implanted with an RNS Neurostimulator or NeuroPace Leads.
* In the investigator's opinion, participant is able to tolerate a neurosurgical procedure.
* Participant with a confirmed diagnosis of idiopathic generalized epilepsy experiencing primary generalized tonic-clonic seizures, with or without myoclonic or absence seizures, consistent with the International League against Epilepsy Revised Classification of Seizures (2017).
* Participant has had 2 or more generalized tonic-clonic seizures during the two month retrospective baseline.
* Participant has had a routine electroencephalogram (EEG) within 2 years prior to enrollment with electroencephalographic features consistent with idiopathic generalized epilepsy; other concomitant anomalies must be explained by adequate past medical history.
* Participant has been on a stable antiseizure medication (ASM) regimen during the two month retrospective baseline and is willing to remain on a stable ASM regimen during the prospective Baseline and throughout the Effectiveness Evaluation Period, if medically possible; rescue benzodiazepine medications for acute seizure clusters are permitted.
* Participant has undergone computed tomography (CT) or magnetic resonance imaging (MRI) within 10 years prior to enrollment that ruled out a progressive cause of epilepsy or an abnormality likely to be associated with focal-onset seizures.
* Participant does not have a vagus nerve stimulator (VNS, LivaNova) or Participant's VNS is OFF during the two month retrospective baseline and participant is willing to keep the VNS off during the study.

Exclusion Criteria:

* Participant is pregnant.
* Participant is participating in a therapeutic investigational drug or other device study.
* Participant is implanted with an electronic medical device that delivers electrical energy to the brain.
* Participant requires procedures that are contraindicated based on current RNS System labeling.
* Participant has been diagnosed with active psychosis, major depression or suicidal ideation in the preceding year. Participants with post-ictal psychiatric symptoms need not be excluded.
* In the opinion of the investigator, the participant has a clinically significant or unstable medical condition (including alcohol and/or drug abuse) or a progressive central nervous system disease.
* Participant has a history of partial-onset seizures or EEG findings within the past 2 years indicative of partial-onset or symptomatic generalized abnormalities.
* Participant has been diagnosed with psychogenic or non-epileptic seizures in the preceding year.
* Participant has experienced unprovoked status epilepticus in the preceding year.
* Participant is taking any anticoagulants.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
12-week post-operative serious device-related adverse event (SADE) rate | 84 days post-implant (12 weeks)
  The primary safety endpoint is the percent of participants with serious device-related adverse events (SADE) at 84 days (12 weeks) post-implant.
Time to second generalized tonic-clonic (GTC) seizure | 9-month Effectiveness Evaluation Period
  The primary effectiveness endpoint is the time to a participant's 2nd GTC seizure (also defined as a GTC-event) during the 9-month Effectiveness Evaluation Period. Across participants, once the 60th GTC-event occurs, the study will have collected the necessary data to assess the primary effectiveness endpoint; all participants will then be unblinded.

SECONDARY OUTCOMES:
Percent change in monthly rate of days with any type of generalized seizure (generalized tonic-clonic, myoclonic, absence) | 9-month Effectiveness Evaluation Period
  The secondary effectiveness endpoint will be the percent change in the monthly rate of days with any type of generalized seizure (generalized tonic-clonic, myoclonic or absence) during the 9-month Effectiveness Evaluation Period compared to baseline.

OTHER OUTCOMES:
Annual event rate of Serious Adverse Device Effects (SADEs) | Implant through 2 years post-implant
  The annual serious adverse device effect (SADE) rate over time in participants implanted with the neurostimulator and/or leads during study participation will be calculated. The SADE event rate is defined as the number of SADEs per implant year.
Annual event rate of Serious Adverse Events (SAEs) of particular relevance | Implant through 2 years post-implant
  The annual rate of serious adverse events (SAEs) of particular relevance (device-related or not) will be calculated over time in participants implanted with the neurostimulator and/or leads during study participation. SAEs of particular relevance include infection, intracranial hemorrhage, suicidality, and cognitive deterioration.
Affective status as assessed by the Beck Depression Inventory | Pre-implant baseline through 2 years post-implant
  Affective status (by summary scores from the Beck Depression Inventory, either the Beck Depression Inventory-II or Beck Youth Inventory-II, depending on age at time of the initial clinic appointment) will be described for the pre-implant baseline, as well as for the post-implant months 6, 12, 18 and 24.
Neuropsychological functioning as assessed by a sub-set of tests in the NIH Toolbox Cognition Battery | Pre-implant baseline through 2 years post-implant
  Neuropsychological functioning as assessed by neuropsychological testing with validated, standardized inventories to assess 3 domains that include attention, memory, and vocabulary (Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, and Picture Vocabulary Test, respectively). These inventories are taken from the NIH Toolbox Cognition Battery and will be described by presenting summary scores for the pre-neurostimulator implant period, as well as for the annual appointments.
Sleep assessment as assessed by sleep habit questionnaires | Pre-implant baseline through 2 years post-implant
  Sleep habits (by summary scores from either the Pittsburgh Sleep Quality Index or Adolescent Sleep Wake Scale, depending on age at time of assessment) will be described for the pre-implant baseline, as well as for the post-implant months 3, 6, 9, 12, 18 and 24.
Health affecting behaviors assessment | Pre-implant baseline through 2 years post-implant
  Health affecting behaviors (by summary scores from either the Millon Behavioral Medicine Diagnostic or Millon Adolescent Clinical Inventory-II, depending on age at time of assessment) will be described for the pre-implant baseline, as well as for the post-implant months 3, 6, 9, 12, 18 and 24.
Percent change in seizure frequency | Blinded Effectiveness Evaluation Period (3 months post-implant up to Time-to-Generalized-Tonic-Clonic-Event)
  The percent change in generalized tonic-clonic seizure frequency will be summarized and reported by medians and responder rates. This variable will be summarized for active and sham groups separately using data collected during the blinded Effectiveness Evaluation Period (3 months post-implant up to Time-to- Generalized-Tonic-Clonic Event).
Quality of life as assessed by the Quality of Life in Epilepsy Inventory | Pre-implant baseline through 2 years post-implant
  Quality of Life in Epilepsy Inventory [by summary scores from the Quality of Life in Epilepsy-AD-48 (validated for ages 12-17 years) or Quality of Life in Epilepsy-31-P (validated for ages 18 and older)], depending on age at time of assessment, will be described for the pre-implant baseline, as well as for the post-implant months 6, 12, 18 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Morrell, MD, Principal Investigator — NeuroPace, Inc.
Locations (23):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Mary Hitchcock Memorial Hospital (Dartmouth), Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - New York University Langone, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No